CLINICAL TRIAL: NCT05447403
Title: Effect of Chewing Gum Combined With Manual Enhanced Instructions by WeChat on the Bowel Preparation Quality for Colonoscopy in Patients With Constipation: a Randomized Controlled Trial
Brief Title: Effect of Chewing Gum and WeChat Enhanced Instructions on the Bowel Preparation Quality in Patients With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Doctor, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XHNKKY-CGCW 1.0
Record Dates: First submitted 2022-03-25; First posted 2022-07-07 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Colonoscopy; Colonic Polyp; Constipation
Keywords: Bowel preparation; Chewing gum; Enhanced instructions; WeChat; Colonoscopy
MeSH Terms: conditions — Colonic Polyps; Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum combined with WeChat enhanced instructions group (Experimental): Patients in the chewing gum and WeChat group are advised to chew one piece of sugarless gum for 20 minutes after drinking each 1 liter PEG. They also receive enhanced instructions via WeChat before two days and one day of colonoscopy to further inform how to chew gum and highlight the importance of adequate bowel preparation.
  Interventions: Other: Chewing gum combined with WeChat enhanced instructions
- Control group (No Intervention): Patients in the control group are guided by regular instructions.

INTERVENTIONS:
Other: Chewing gum combined with WeChat enhanced instructions — Patients in the chewing gum and WeChat group are advised to chew one piece of sugarless gum for 20 minutes after drinking each 1 liter PEG. They also receive enhanced instructions via WeChat before two days and one day of colonoscopy to further inform how to chew gum and highlight the importance of adequate bowel preparation.
  Arms: Chewing gum combined with WeChat enhanced instructions group

SUMMARY:
Patients with constipation are more likely to have poor bowel preparation quality due to slow gut motility and poor emptying ability. Gum chewing, as a proxy of sham feeding, is a very simple way used to accelerate gut motility. And a previous study found that enhanced instructions by WeChat could improve bowel preparation quality. Thus, investigators conducted a single-center randomized controlled trial to explore the effect of chewing gum combined with manual enhanced instructions by WeChat on the bowel preparation quality for colonoscopy in patients with constipation.

DETAILED DESCRIPTION:
In this randomized controlled trial, consecutive outpatients with constipation for colonoscopy are screened and then randomized into two groups. All enrolled patients will receive 3 liter polyethylene glycol (PEG) for bowel preparation. Patients in the chewing gum and WeChat group (n = 75) are further advised to chew one piece of sugarless gum for 20 minutes after drinking each 1 liter PEG; additionally, they will receive enhanced instructions via WeChat before two days and one day of colonoscopy to further inform how to chew gum and highlight the importance of adequate bowel preparation. Patients in the control group (n = 75) are guided by regular instructions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing colonoscopy at the Department of Gastroenterology of the General Hospital of Northern Theater Command.
2. Patients aged ≥18 years, no gender limitation.
3. Patients who sign informed consent.
4. Patients who are diagnosed with constipation.

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Patients who are allergic to polyethylene glycol.
3. Patients who are suspected with intestinal obstruction, stenosis or perforation.
4. Patients with mental illness.
5. Patients with serious heart, brain, liver, and kidney diseases.
6. Patients who use WeChat unconditionally by themselves or their family members.
7. Patients who are allergic to chewing gum related ingredients.
8. Patients with the history of colorectal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality | During colonoscopy procedure, an average of 30 minutes
  Bowel preparation quality is evaluated by the Boston bowel preparation scale (BBPS) score:
  Segment score 0: unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared.
  Segment score 1: portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid.
  Segment score 2: minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well.
  Segment score 3: entire mucosa of colon segment seen well with no residual staining, small fragments of stool and/or opaque liquid.

SECONDARY OUTCOMES:
The number of polyp and/or adenoma | During colonoscopy procedure, an average of 30 minutes
  The number of polyp and/or adenoma is defined as the number of adenoma/polyp detected during colonoscopy.
Polyp and/or adenoma detection rate | During colonoscopy procedure, an average of 30 minutes
  Polyp and/or adenoma detection rate (PDR/ADR) is defined as the proportion of patients with at least one histologically confirmed adenoma/polyp detected during colonoscopy.
Adverse events | During colonoscopy procedure, an average of 30 minutes
  Adverse events are defined as the occurrence of gastrointestinal symptoms during bowel preparation, including nausea, vomiting, abdominal pain, and bloating.
Cecal intubation time | During colonoscopy procedure, an average of 30 minutes
  Cecal intubation time (CIT) is defined as the time from the insertion of the colonoscope tip into the anal verge until reaching the cecal base or cecal end.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, MD, Principal Investigator — The General Hospital of Northern Theater Command; Cong Gao, MS, Principal Investigator — The General Hospital of Northern Theater Command; Fei Gao, MD, Principal Investigator — The General Hospital of Northern Theater Command
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

REFERENCES:
- [Background] Lu J, Cao Q, Wang X, Pu J, Peng X. Application of Oral Lactulose in Combination With Polyethylene Glycol Electrolyte Powder for Colonoscopy Bowel Preparation in Patients With Constipation. Am J Ther. 2016 Jul-Aug;23(4):e1020-4. doi: 10.1097/MJT.0000000000000351. PMID 26658804
- [Background] Lee J, Lee E, Kim Y, Kim E, Lee Y. Effects of gum chewing on abdominal discomfort, nausea, vomiting and intake adherence to polyethylene glycol solution of patients in colonoscopy preparation. J Clin Nurs. 2016 Feb;25(3-4):518-25. doi: 10.1111/jocn.13086. PMID 26818376
- [Background] Wang SL, Wang Q, Yao J, Zhao SB, Wang LS, Li ZS, Bai Y. Effect of WeChat and short message service on bowel preparation: an endoscopist-blinded, randomized controlled trial. Eur J Gastroenterol Hepatol. 2019 Feb;31(2):170-177. doi: 10.1097/MEG.0000000000001303. PMID 30418256